CLINICAL TRIAL: NCT00150995
Title: A Phase II Trail of Tetrathiomolybdate in Patients With Hormone Refractory Prostate Cancer
Brief Title: Tetrathiomolybdate in Hormone Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9962
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tetrathiomolybdate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tetrathiomolybdate (Experimental): Patients will be started on a dose of 60mg Tetrathiomolybdate at bedtime and 40mg 3 times per day.
  Interventions: Drug: Tetrathiomolybdate

INTERVENTIONS:
Drug: Tetrathiomolybdate

SUMMARY:
Purpose: The aim of this clinical trail is to evaluate Tetrathiomolybdate (TM) in the treatment of hormone refractory prostate cancer.

DETAILED DESCRIPTION:
Tetrathiomolybdate or TM, a drug developed for Wilson's Disease, removes copper from the bloodstream. Copper is a key factor in angiogenesis (blood vessel growth)- a process that occurs normally in the body but becomes uncontrolled in cancerous cells. Tetrathiomolybdate essentially wages war against copper, which serves to choke off tumor growth. Realizing the key role of copper in angiogenesis, researchers have begun exploring treatment with Tetrathiomolybdate for different types of cancers. This clinical trial will evaluate the effectiveness of Tetrathiomolybdate in the treatment of patients with hormone refractory prostate cancer. Hormone refractory prostate cancer refers to advanced disease in which the patient no longer responding to conventional hormonal treatment.

ELIGIBILITY:
Inclusion:

* Patients must have histologic diagnosis of adenocarcinoma of the prostate with progression following hormonal therapy and antiandrogen withdrawal.
* Patients must have minimal disease (defined as bone metastasis or visceral disease with no impairment of organ function or pain severe enough to require narcotics for control).
* Adequate bone marrow and renal function
* ECOG (Eastern Cooperative Oncology Group) score of 0 or 1 (a measure of general well being where 1 represents asymptomatic and 5 represents death)
* Life expectancy of at least 16 weeks
* Must have completed radiation more than 4 weeks prior to registration and must have a rising PSA (Prostate Specific Antigen) and lesion outside of the radiation field

Exclusion:

* Patients with an elevated PSA as the only evidence of disease
* Clinical evidence of spinal cord compression
* History of prior malignancy within the past 5 years (with the exception of in situ carcinoma of any site or nonmelanoma skin cancer)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2001-05; Primary Completion 2003-10 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Time to Progression | 12 weeks
  To determine the time to progression of prostate cancer in patients with androgen-independent prostate cancer treated with tetrathiomolybdate. Disease progression is defined as at least a 20% increase in the sum of the longest diameter of the target lesions. For disease evaluable only by bone scan, the appearance of new lesions was considered evidence of progression. The development of pain in an existing lesion requiring institution of palliative radiotherapy or prescription narcotics was also considered evidence of progression.

CONTACTS AND LOCATIONS:
Overall Officials: David C. Smith, MD, Principal Investigator — The University of Michigan Comprehensive Cancer Center
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States